CLINICAL TRIAL: NCT05572593
Title: Utility of Pharmacogenomic Testing in Patients With Gastrointestinal Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Adil Bharucha, MBBS, MD, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 16-008401
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2022-10-07 (Actual); Status verified 2022-10

CONDITIONS: Gastrointestinal Diseases
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Pharmacogenomic Testing; Genetic Testing

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Group (Experimental): Subjects treating physician will receive PGx results to facilitate clinical decisions
  Interventions: Genetic: Pharmacogenomics (PGx) genetic testing
- Unguided Group (Active Comparator): Subjects treating physician will be blinded to PGx results and will receive standard medical care
  Interventions: Genetic: Pharmacogenomics (PGx) genetic testing

INTERVENTIONS:
Genetic: Pharmacogenomics (PGx) genetic testing — A buccal swab to collect cells from the inside the cheek

SUMMARY:
Researchers are trying to learn more about how individuals break down and process specific medications based on their genes. Pharmacogenomics (PGx) is a new, specialized field within individualized medicine. PGx is the study of how genes may affect the body's response to, and interaction with, some prescription medications. Genes carry information that determines things such as eye color and blood type. Genes can also influence how individuals process and respond to medications. Depending on genetic make-up, some medications may work faster or slower or produce fewer side effects.

ELIGIBILITY:
Inclusion Criteria

* Rome IV criteria for functional nausea and vomiting disorders (chronic nausea vomiting syndrome, cyclic vomiting syndrome), abdominal bloating/distention, dyspepsia, irritable bowel syndrome, chronic abdominal pain, functional diarrhea, or chronic constipation.
* On 1 or more medications identified in Appendix 1 on a daily basis for at least six months.
* Symptoms of moderate or severe severity on either of these 2 instruments: For IBS-SSS, use moderate (175-300) or severe (> 300) IBS. For FD - Score ≥ 3 for any symptom on Nepean Dyspepsia Index.
* No prior pharmacogenomics assessment.
* Willingness to adjust medications based upon results of PGX testing.
* Patients must understand and provide written informed consent and HIPAA authorization prior to initiation of any study-specific procedures.
* Patients must have the ability to complete questionnaires by themselves or with assistance.

Exclusion Criteria:

* Patients who decline to be evaluated by a mental health professional during their evaluation.
* Rumination syndrome, cannabinoid hyperemesis syndrome, patients with a significant GI disease process (e.g., intestinal pseudo-obstruction, severe gastroparesis, megacolon) which, in the opinion of the investigator, is likely irreversible.
* Patients who, in the opinion of the investigator, are likely to undergo another major therapeutic intervention during the next 6 months (e.g., surgery or pelvic floor retraining by biofeedback therapy). However, other changes (e.g., medications) will not preclude participation in the study.
* Patients with any of the following per history, and review of medical record prior to study entry: any psychotic disorders, bipolar disorders, or major cognitive disorders; any active substance use disorders, other than tobacco; currently active suicidal ideation; current treatment with electroconvulsive therapy (ECT) or repetitive transcranial magnetic stimulation (rTMS); discharge from a psychiatric inpatient hospital or intensive psychiatric outpatient program within 6 weeks prior to GI consultation.
* Patients who are unwilling or cannot, for any reason, adjust their medications.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Number of subjects to have clinical management changes based on PGx results | 3 months
  Number of subjects that pharmacogenomic (PGx) results guided the clinical management of gastrointestinal disorders
Change in Irritable Bowel Syndrome (IBS) severity | Baseline, 3 months. 6 months
  Measured using the self-reported IBS severity scoring system (IBS-SSS) Questionnaire; 500 point continuous scale: 0= no symptoms to 500=maximum severity
Change in Irritable Bowel Syndrome Quality of Life | Baseline, 3 months. 6 months
  Measured using the self-reported Irritable Bowel Syndrome Quality of Life (IBS-QOL) survey; score ranges from 0 (poor QOL) to 100 (maximum QOL)
Change in symptom severity with dyspepsia | Baseline, 3 months. 6 months
  Measured using the self-reported Nepean Dyspepsia Index (NDI) questionnaire which consists of a symptom checklist that measures frequency (0-4), intensity (0-5) and bothersomeness (0-4) of 15 upper gastrointestinal symptoms. The average score for each symptom is derived by averaging scores for frequency, intensity, and bothersomeness. Scores of 3 respectively represent a frequency of 9 to 12 days/week, moderate intensity, and a bothersomeness of "quite a bit".

SECONDARY OUTCOMES:
Change in anxiety | Baseline, 3 months, 6 months
  Measured using the self-reported Generalized Anxiety Disorder-7 (GAD-7) questionnaire; score range 0-21 points, higher scores indicate worse symptoms
Change in Patient Health Questionnaire Score | Baseline, 3 months, 6 months
  Measured using the self-reported Patient Health Questionnaire (PHQ-9); score range 0-27 points, higher scores indicate worse symptoms
Change in general well-being | Baseline, 3 months, 6 months
  Measured using the self-reported Global Wellbeing Likert scale; subjects asked to rate their general health perception on a scale range of 1=Excellent, 2=Very Good, 3=Good, 4=Fair, 5=Poor
Change in Pain score | Baseline, 3 months, 6 months
  Measured using the self-reported McGill Pain score; score range 0-78; higher scores indicate worse pain

CONTACTS AND LOCATIONS:
Overall Officials: Adil Bharucha, MBBS, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials